CLINICAL TRIAL: NCT02344797
Title: Prevention of Myocardial Injury by Remote Ischemic Preconditioning in Emergent or Urgent Non-cardiac Surgery: a Randomized Clinical Trial
Brief Title: Prevention of Myocardial Injury in Non-cardiac Surgery
Acronym: PIXIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Sarah Victoria Ekeløf Busch, MD, Ph.d. student, Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SBpixie
Record Dates: First submitted 2015-01-13; First posted 2015-01-26 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Myocardial Injury; Myocardial Infarction
Keywords: Perioperative; Postoperative Complications/prevention & control
MeSH Terms: conditions — Myocardial Infarction; Postoperative Complications

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Remote ischemic preconditioning, 4 cycles of 5 minutes ischemia and 5 minutes reperfusion of the forearm before surgery.
  Interventions: Procedure: Remote ischemic preconditioning
- Control (No Intervention)

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — The remote ischemic preconditioning procedure is carried out immediately after the induction of regional or general anesthesia. The blood pressure cuff is placed on the upper limb. The cuff is inflated to 200 mmHg resulting in a total occlusion of the blood flow to the limb. After 5 minutes of ischemia the cuff is deflated and the limb is reperfused for 5 minutes. The procedure is carried out 4 times in a row. For patients with systolic blood pressures >185 mmHg, the cuff will be inflated to at least 15 mmHg above the patient's systolic blood pressure.
  Arms: Intervention

SUMMARY:
Worldwide, more than 200 million patients have major non-cardiac surgery annually and a significant proportion of these patients suffer major cardiovascular complications (e.g. nonfatal myocardial infarction, cardiac arrest, vascular death) within 30 days of their surgery. Perioperative myocardial infarction is the most common cardiovascular complication and recent clinical studies have shown that even minor myocardial injury in relation to non-cardiac surgery is associated with 30-day mortality.

Remote ischemic preconditioning is a procedure, which protects remote tissues and organs e.g. against ischemia-reperfusion injury. Cycles of forearm or leg ischemia and reperfusion by the inflation of a blood-pressure cuff for brief periods are the preferred method.The aim of this interventional clinical study is to determine whether remote ischemic preconditioning can reduce markers of myocardial injury in emergent or urgent non-cardiac surgery.

DETAILED DESCRIPTION:
Patients with a hip fracture will be included in the study. The patients will be randomized to remote ischemic preconditioning or control (no intervention). The remote ischemic preconditioning procedure is carried out immediately after the induction of regional or general anesthesia. The blood pressure cuff is placed on the upper limb. The cuff is inflated to 200 mmHg resulting in a total occlusion of the blood flow to the limb. After 5 minutes of ischemia the cuff is deflated and the limb is reperfused for 5 minutes. The procedure is carried out 4 times in a row. For patients with systolic blood pressures >185 mmHg, the cuff will be inflated to at least 15 mmHg above the patient's systolic blood pressure.

The primary outcome is myocardial injury in noncardiac surgery within day 4 postoperatively.

We expect 15% of the patients in the placebo group to suffer myocardial injury while the incidence of myocardial injury is expected to be reduced to 7% in the intervention group. Type I error is set at 5% and type II error is set at 20%. In total 2 x 264 patients need to be included based on this power calculation. We will include patients until we have a total of 2 x 270 patients for evaluation (per-protocol).

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 45 years undergoing in-hospital hip fracture surgery
* undergoing emergent or urgent surgery (i.e. emergent or urgent visitation to the Department of Orthopedic Surgery)
* fulfil 1 or more of the following 4 inclusion criteria, which are all determined during the conversation with the patient:

  1. Ischemic heart disease, defined by any of the following criteria A. angina pectoris B. prior myocardial infarction C. prior percutaneous coronary intervention D. prior coronary artery bypass graft
  2. Peripheral arterial disease, defined by any of the following criteria A. intermittent claudication B. reduced peripheral arterial blood flow C. prior vascular surgery due to peripheral arterial disease
  3. Prior stroke OR
  4. any 1 of 7 risk criteria A. age ≥70 years; B. congestive heart failure C. prior transient ischemic attack; D. diabetes and currently taking an oral hypoglycemic agent or insulin E. hypertension G. preoperative serum creatinine >175 µmol/L (>2.0 mg/dl) H. smoking within 2 years of surgery

Exclusion Criteria:

* History of peripheral arterial disease affecting both upper limbs
* Renal failure with eGRF<30ml/min/1.73m2
* Cardiogenic shock or cardiac arrest during the current hospital admission
* Reoperation after elective surgery carried out during the current hospital admission
* Not capable of giving informed consent after oral and written information
* Other conditions that prevent the performance of remote ischemic preconditioning.
* Previously included in this trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2015-02-07; Primary Completion 2017-09 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Number of patients with myocardial injury in non-cardiac surgery | during surgery or the first 4 days after surgery

SECONDARY OUTCOMES:
Peak plasma TnI and total TnI release (area under the curve) | during surgery or the first 4 days after surgery
Endothelial dysfunction (reactive hyperemia index) | 24 hours after surgery
  Assessed by EndoPat
Perioperative myocardial infarction | 30 days, one year and 5 years after surgery
Major adverse cardiovascular events | 30 days, one year and 5 years after surgery
Length of postoperative hospital stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
Length of intensive care unit stay | participants will be followed for the duration of hospital stay, an expected average of 10 days
All-cause mortality | 30 days, one year and 5 years after surgery
Biomarkers of coagulation | preoperatively, 2 hours after incision, and on days 1 and 2 after surgery
Plasma N-terminal Pro-Brain Natriuretic Peptide | Preoperative and day 1
  Plasma N-terminal Pro-Brain Natriuretic Peptide (NT-proBNP) before surgery and at day 1 after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Busch, MD, Principal Investigator — Department of Surgery, Koge Hospital, Denmark
Locations (3):
- Denmark (3):
  - Depertment of Orthopedic Surgery, Holstebro Hospital, Holstebro, Central Jutland
  - Department of Anesthesia, Herlev Hospital, Herlev, Region H
  - Department of Surgery, Koge Hospital, Køge

REFERENCES:
- [Derived] Wahlstrom KL, Ekeloef S, Gogenur I, Munster AB. Myocardial injury after non-cardiac surgery and per operative fibrin metabolism in patients undergoing hip-fracture surgery: an observational study. Scand J Clin Lab Invest. 2023 Sep;83(5):299-308. doi: 10.1080/00365513.2023.2220970. Epub 2023 Aug 16. PMID 37584362
- [Derived] Ekeloef S, Koyuncu S, Holst-Knudsen J, Gundel O, Meyhoff CS, Homilius M, Stilling M, Ekeloef P, Munster AMB, Mathiesen O, Gogenur I. Cardiovascular events in patients undergoing hip fracture surgery treated with remote ischaemic preconditioning: 1-year follow-up of a randomised clinical trial. Anaesthesia. 2021 Aug;76(8):1042-1050. doi: 10.1111/anae.15357. Epub 2021 Jan 13. PMID 33440017
- [Derived] Ekeloef S, Homilius M, Stilling M, Ekeloef P, Koyuncu S, Munster AB, Meyhoff CS, Gundel O, Holst-Knudsen J, Mathiesen O, Gogenur I. The effect of remote ischaemic preconditioning on myocardial injury in emergency hip fracture surgery (PIXIE trial): phase II randomised clinical trial. BMJ. 2019 Dec 4;367:l6395. doi: 10.1136/bmj.l6395. PMID 31801725

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/97/NCT02344797/Prot_SAP_000.pdf